CLINICAL TRIAL: NCT00972764
Title: Laryngomalacia No Longer An Ambiguity
Status: Completed | Type: Observational
Sponsor: Boushahri Clinic Medical Center (Other)
Responsible Party: Principal Investigator, Mohamed Said El-Sayed, Professor, Boushahri Clinic Medical Center
Other Study IDs: 461956 (BoushahriCMC)
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Laryngomalacia
Keywords: Laryngomalacia; Factors Associated or Predisposing
MeSH Terms: conditions — Laryngomalacia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control
- Laryngomalacia Cases

SUMMARY:
The purpose of this study is to expose some of the factors that may be associated or predisposing to development of laryngomalacia.

DETAILED DESCRIPTION:
Laryngomalacia is the most common congenital malformation of the larynx and it is a self-limited disorder. It is the most common cause of stridor in newborns and infants. It results from an abnormal prolapse of supraglottic structures during inspiration. Despite its widespread prevalence, the etiology of laryngomalacia is unclear. Most infants will squeaky but otherwise well. Although affected patients do not exhibit much in the way of other physical symptoms, the unusual voice is worrisome to their parents.

ELIGIBILITY:
Inclusion Criteria:

* Babies delivered with laryngomalacia with ≥ 37 weeks of gestation
* Delivered with birth weights ≥ 2.5 kg
* No history of natal or post-natal complications
* From the same community

Exclusion Criteria:

* Pre-term babies
* History of natal or post-natal complications

Ages: 14 Days to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Primary care clinics
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2006-01; Primary Completion 2008-07 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S EL-Sayed, MBBCh,MSc,MD, Principal Investigator — New Children's Hospital, Cairo University
Locations (1):
- Boushahri Clinic Medical Center, Kuwait City, P.O.Box :698 Salmiya, Kuwait